CLINICAL TRIAL: NCT05992987
Title: Assessment of Serum Levels of Adenosine Deaminase and Immunoglobulin E in Patients With Chronic Spontaneous Urticaria
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed, Resident physician at Dermatology department, Sohag University, Sohag University
Other Study IDs: Soh-Med-23-07-12MS
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: chronic spontaneous urticaria; adenosine deaminase; immunoglobulin E
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- CSU group: Adult patients complaining of chronic spontaneous urticaria (CSU)
  Interventions: Diagnostic Test: Adenosine deaminase serum level; Diagnostic Test: IgE antibodies serum level
- Control group: A group of age and sex-matched healthy controls (blood donors).
  Interventions: Diagnostic Test: Adenosine deaminase serum level; Diagnostic Test: IgE antibodies serum level

INTERVENTIONS:
Diagnostic Test: Adenosine deaminase serum level — Adenosine deaminase will be measured by enzymatic (clorometric / kinetic) method (Diazyme laboratories, San Diego, California, USA).
Diagnostic Test: IgE antibodies serum level — Level of IgE will be measured by electrochemiluminesence immunoassay (ECLIA, automatic cobase immunoassay, Roche Diagnostics GmbH, Mannheim, USA).

SUMMARY:
adenosine deaminase activity (ADA) has been reported to be elevated in various diseases such as psoriasis, acne and juvenile idiopathic arthritis. There is no previous studies that assessed ADA in chronic spontaneous urticaria (CSU) .

ELIGIBILITY:
Inclusion Criteria:

* adult patients complaining of CSU and a group of age and sex-matched healthy controls (blood donors).

Exclusion Criteria:

* Pregnancy and lactation.
* Patients with systemic diseases, especially those with autoimmune diseases and infections.
* Patients with skin diseases.
* Patients on medications such as antibiotics, nonsteroidal anti-inflammatory drugs, angiotensin-converting enzyme inhibitors, anticonvulsants, penicillin, and combined oral contraceptives.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Settings: Dermatology outpatient clinics and Central Research Lab at Sohag University.
  Study population: The study will include adult patients complaining of CSU and a group of age and sex-matched healthy controls (blood donors).
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Serum level of adenosine deaminase | 3 months
  Difference in serum level of adenosine deaminase between CSU group and control group
Serum level of IgE | 3 months
  Difference in serum level of IgE between CSU group and control group

CONTACTS AND LOCATIONS:
Overall Officials: Ramadan Saleh, MD, Study Director — Sohag University

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon request to the study director
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available after study due for unlimited period of time.
Access Criteria: IPD will be shared upon request by the study director. Patients' names will be anonymous.